CLINICAL TRIAL: NCT01732835
Title: The HAART 300 Annuloplasty Ring Extended Safety and Performance Trial Used in Surgical Repair of the Aortic Valve
Brief Title: The HAART 300 Annuloplasty Ring Trial Extended Safety and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biostable Science & Engineering (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-01-022
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Aortic Insufficiency
Keywords: Aortic Insufficiency (AI) Aortic Regurgitation (AR)
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HAART 300 Annuloplasty Device (Experimental): Implantation of HAART 300 Annuloplasty Device for aortic valve repair
  Interventions: Device: HAART 300 Annuloplasty Device

INTERVENTIONS:
Device: HAART 300 Annuloplasty Device — Implantation of HAART 300 Annuloplasty Device for aortic valve repair

SUMMARY:
This investigation is a prospective, non-randomized, multi-center trial to evaluate the extended safety and performance of the HAART model 300 annuloplasty ring when used to surgically repair the aortic valve using a 3-D intra-annular mounting frame.

DETAILED DESCRIPTION:
Aortic Regurgitation, (also known as Aortic Insufficiency; AI), is the failure of the aortic valve to close completely during diastole which causes blood to flow from the aorta back into the left ventricle. Aortic Regurgitation (AR) is a frequent cause of both disability and death due to congestive heart failure, primarily in individuals forty or older, but can also occur in younger populations.

Traditionally management of aortic regurgitation has been by aortic valve replacement, however, as has been observed in patients who have had mitral valve repair, the option of maintaining ones native aortic valve versus a replacement, either bioprosthetic or mechanical, can have added multiple benefits. The advantage of repair is the avoidance of prosthetic valve-related complications with bioprosthetic valves over 10-15 years or the need for anticoagulation with mechanical valves and the related problems of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older
* Subject has tri-leaflet aortic valve morphology
* Subject has documented aortic valve disease which may or may not include:

  1. aortic valve insufficiency
  2. aortic root pathology
  3. pathology of the ascending aorta
  4. patients with associated stable one or two vessel coronary disease requiring concomitant coronary bypass
* Subject is willing to comply with specified follow-up evaluations, including transesophageal echocardiography (TEE) if there are inadequate images by transthoracic echocardiography (TTE) to assess the aortic valve
* Subject has reviewed and signed the written informed consent form
* Subject agrees to return for all follow-up evaluations for the duration of the study (i.e.,. geographically stable)

Exclusion Criteria:

* The subject has pre-existing valve prosthesis in the aortic position
* The subject's aortic valve morphology is not tri-leaflet
* The subject has active endocarditis
* Heavily calcified valves
* The subject has mixed stenosis and regurgitation of the aortic valve with predominant stenosis
* Leukopenia
* Acute anemia (Hb < 9mg%)
* Platelet count <100,000 cell/mm3
* Need for emergency surgery for any reason
* History of bleeding diathesis or coagulopathy or the subject refuses blood transfusions
* Active infection requiring antibiotic therapy (if temporary illness, subjects may enroll 4 weeks after discontinuation of antibiotics)
* Subjects in whom transesophageal echocardiography (TEE) is contraindicated
* Low Ejection Fraction (EF) EF < 35%
* Life expectancy < 1 year
* The subject is or will be participating in a concomitant research study of an investigational product or has participated in such a study within the 30 days prior to screening
* The subject is a minor, an illicit drug user, alcohol abuser, prisoner, institutionalized, or is unable to give informed consent
* The subject is pregnant or lactating
* Recent (within 6 months) cerebrovascular accident (CVA) or a transient ischemic attack (TIA)
* Myocardial Infarction (MI) within one month of trial inclusion
* The subject has a known intolerance to titanium or polyester
* The subject has documented unstable or > 2 vessel coronary disease
* The subject requires additional valve replacement or valve repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominico Mazzitelli, MD, Principal Investigator — Munchen Heart Center
Locations (8):
- Institute of Clinical and Experimental Medicine, Prague, Czechia
- Germany (7):
  - German Heart Center, Berlin
  - Uniklinik Köln, Cologne
  - Klinik für Herz und Gefässchirurgie, Freiburg im Breisgau
  - Klinik und Poliklinik für Herz- und Gefäßchirurgie, Hamburg
  - Hannover Medical School (MHH), Hanover
  - Munchen Heart Center, München
  - Klinikum Nürnberg Süd, Nuremberg

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: 6-month Primary Endpoint
Arm/Group | HAART 300 Annuloplasty Device
Started | 68
Completed | 44
Not Completed | 24
Not completed — Did not receive device | 19
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 3
Period: 2-year Extended Follow-up
Arm/Group | HAART 300 Annuloplasty Device
Started | 44
Completed | 39
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Participants with implanted device
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 32
Region of Enrollment [Number; unit: participants]
  Czech Republic | 5
  Germany | 44
Aortic Insufficiency [Number; unit: participants] — Grade assigned to degree of aortic regurgitation determined by core laboratory analysis of echocardiogram: 0=None/trace, 1+=Mild, 2+=Moderate, 3+=Moderate-to-Severe, 4+=Severe
  participants
    0 | 0
    1+ | 3
    2+ | 10
    3+ | 18
    4+ | 12
    Not evaluable | 6
New York Heart Association (NYHA) Functional Capacity [Number; unit: participants] — Four classes describing the effect of cardiac disease on physical activity: Class I - disease does not limit activity; Class II - slight limitation; Class III - marked imitation; Class IV - inability to carry out any physical activity without discomfort
  participants
    I | 11
    II | 25
    III | 13
    IV | 0
Peak gradient [Mean (Standard Deviation); unit: mm Hg] — Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  mm Hg
    number analyzed (Participants) | 43
    (all) | 11.1 (4.7)
Mean gradient [Mean (Standard Deviation); unit: mm Hg] — Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  mm Hg
    number analyzed (Participants) | 43
    (all) | 5.5 (2.4)
Left ventricular (LV) mass [Mean (Standard Deviation); unit: g] — Left ventricular mass. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  g
    number analyzed (Participants) | 39
    (all) | 244.1 (85.2)
Left ventricular internal dimension (LVID) diastole [Mean (Standard Deviation); unit: cm] — Left ventricular internal dimension. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  cm
    number analyzed (Participants) | 40
    (all) | 5.50 (0.86)
LVID systole [Mean (Standard Deviation); unit: cm] — Left ventricular internal dimension. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  cm
    number analyzed (Participants) | 35
    (all) | 4.02 (0.83)
LV diastolic volume [Mean (Standard Deviation); unit: ml] — Left ventricular diastolic volume. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  ml
    number analyzed (Participants) | 27
    (all) | 155.3 (63.3)
LV systolic volume [Mean (Standard Deviation); unit: ml] — Left ventricular systolic volume. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  ml
    number analyzed (Participants) | 28
    (all) | 76.5 (37.7)
Left ventricular ejection fraction (LVEF) [Mean (Standard Deviation); unit: %] — Left ventricular ejection fraction. Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  %
    number analyzed (Participants) | 27
    (all) | 54.2 (4.4)
Cardiac output [Mean (Standard Deviation); unit: l/min] — Echocardiographic parameter determined by core laboratory. Population: Participants with an echocardiogram evaluable for this measure.
  l/min
    number analyzed (Participants) | 32
    (all) | 6.20 (2.17)
Cardiac index [Mean (Standard Deviation); unit: l/min/m^2] — Cardiac index is the cardiac output divided by body surface area. Population: Participants with an echocardiogram evaluable for this measure.
  l/min/m^2
    number analyzed (Participants) | 32
    (all) | 3.16 (1.11)

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Outcome Measure: Survival Defined as Survival Free From All Cause Death at 6 Months Postprocedure
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 49
percentage of participants | 100 [92.8 to 100]

2. Primary Outcome: Primary Efficacy Outcome Measure: Aortic Insufficiency (AI) at 6 Months
Description: Assessed by transthoracic echocardiography (TTE) and graded as None/Trace (0), Mild (1+), Moderate (2+), Moderate-to-Severe (3+), or Severe (4+)
Time Frame: 6 months
Population: Participants with an echocardiogram evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 41
participants
  0 | 11
  1+ | 21
  2+ | 7
  3+ | 2
  4+ | 0

3. Secondary Outcome: Implant Procedure Success
Description: Success is defined as the absence of specified adverse events evaluated through discharge or 14 days after the procedure: - Aortic annular dissection, rupture, or leaflet damage - Mitral valve impingement due to implant - implant dehiscence/migration into aorta - implant dehiscence/migration into left ventricle - Hemodynamics requiring intervention - Other adverse event resulting in reoperation, explantation, or permanent disability.
Time Frame: discharge or 14 days postprocedure, whichever comes first
Measure: Number (95% Confidence Interval); unit: percentage of implant procedures
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 49
percentage of implant procedures | 95.9 [86.0 to 99.5]

4. Secondary Outcome: Actuarial Freedom From Clinical Cardiovascular Events
Description: Freedom from specified clinical cardiovascular events at 6 months postprocedure: - Device-related mortality - Complete heart block - Structural device failure - Endocarditis - Periprosthetic leak or dehiscence - Thromboembolism - Bleeding Event - Native Valve Deterioration - Valve Thrombosis - Hemolysis - Reoperation and explant at 6 months
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 49
percentage of participants | 89.6 [80.9 to 98.4]

5. Secondary Outcome: Survival Defined as Survival Free From All Cause Death at 2 Years Postprocedure
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 49
percentage of participants | 97.6 [83.9 to 99.7]

6. Secondary Outcome: Aortic Insufficiency (AI) at 2 Years
Description: as for outcome 2
Time Frame: 2 years
Population: Participants with an echocardiogram evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 37
participants
  0 | 2
  1+ | 25
  2+ | 10
  3+ | 0
  4+ | 0

7. Secondary Outcome: New York Heart Association (NYHA) Functional Capacity Classification at 6 Months
Description: Four classes describing the effect of cardiac disease on physical activity: Class I - disease does not limit activity; Class II - slight limitation; Class III - marked limitation; Class IV - inability to carry out any physical activity without discomfort
Time Frame: 6 months
Population: Participants with an evaluation of this measure.
Measure: Number; unit: participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 43
participants
  I | 30
  II | 13
  III | 0
  IV | 0

8. Secondary Outcome: New York Heart Association (NYHA) Functional Capacity Classification at 2 Years
Description: as for outcome 7
Time Frame: 2 years
Population: Participants with an evaluation of this measure.
Measure: Number; unit: participants
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 38
participants
  I | 28
  II | 9
  III | 1
  IV | 0

9. Secondary Outcome: Peak Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 36
mm Hg | 5.3 (6.7)

10. Secondary Outcome: Peak Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 34
mm Hg | 5.9 (10.7)

11. Secondary Outcome: Mean Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 36
mm Hg | 2.6 (3.7)

12. Secondary Outcome: Mean Gradient - Change From Baseline
Description: Transthoracic echocardiography parameter
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 34
mm Hg | 3.1 (5.3)

13. Secondary Outcome: LV Mass - Change From Baseline
Description: Left ventricular mass. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 29
g | -26.5 (60.0)

14. Secondary Outcome: LV Mass - Change From Baseline
Description: Left ventricular mass. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 24
g | -27.4 (60.8)

15. Secondary Outcome: LVID Diastole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 30
cm | -0.48 (0.71)

16. Secondary Outcome: LVID Diastole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 24
cm | -0.22 (0.65)

17. Secondary Outcome: LVID Systole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 25
cm | -0.48 (0.71)

18. Secondary Outcome: LVID Systole - Change From Baseline
Description: Left ventricular internal dimension. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 17
cm | -0.22 (0.84)

19. Secondary Outcome: LV Diastolic Volume - Change From Baseline
Description: Left ventricular diastolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
ml | -21.8 (49.2)

20. Secondary Outcome: LV Diastolic Volume - Change From Baseline
Description: Left ventricular diastolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 18
ml | -19.9 (53.0)

21. Secondary Outcome: LV Systolic Volume - Change From Baseline
Description: Left ventricular systolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 17
ml | -17.5 (30.2)

22. Secondary Outcome: LV Systolic Volume - Change From Baseline
Description: Left ventricular systolic volume. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 19
ml | -11.1 (29.1)

23. Secondary Outcome: LVEF - Change From Baseline
Description: Left ventricular ejection fraction. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Error); unit: percentage of blood volume
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 16
percentage of blood volume | 2.49 (7.65)

24. Secondary Outcome: LVEF - Change From Baseline
Description: Left ventricular ejection fraction. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 18
percentage of blood volume | 0.37 (7.19)

25. Secondary Outcome: Cardiac Output - Change From Baseline
Description: Stroke volume x heart rate. Transthoracic echocardiography parameter.
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 22
l/min | -1.15 (1.66)

26. Secondary Outcome: Cardiac Output - Change From Baseline
Description: Stroke volume x heart rate. Transthoracic echocardiography parameter.
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 20
l/min | -0.50 (2.20)

27. Secondary Outcome: Cardiac Index - Change From Baseline
Description: Hemodynamic parameter computed as cardiac output divided by body surface area
Time Frame: Baseline and 6 months
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 6 months.
Measure: Mean (Standard Deviation); unit: l/min/m^2
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 22
l/min/m^2 | -0.60 (0.85)

28. Secondary Outcome: Cardiac Index - Change From Baseline
Description: Hemodynamic parameter computed as cardiac output divided by body surface area
Time Frame: Baseline and 2 years
Population: Participants with an echocardiogram evaluable for this measure at baseline and at 2 years.
Measure: Mean (Standard Deviation); unit: l/min/m^2
Arm/Group | HAART 300 Annuloplasty Device
Number analyzed (Participants) | 20
l/min/m^2 | -0.26 (1.07)

ADVERSE EVENTS:
Time Frame: Through 2 years for the 49 participants receiving the implant
Arm/Group | HAART 300 Annuloplasty Device
Serious Adverse Events (participants affected / at risk) | 23/49
Other Adverse Events (participants affected / at risk) | 38/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAART 300 Annuloplasty Device (N=49)
angina pectoris (Cardiac disorders) | 1 (1)
aortic insufficiency (Cardiac disorders) | 5 (5)
arrhythmia (Cardiac disorders) | 4 (5)
cardiac decompensation (Cardiac disorders) | 1 (1)
pericardial effusion (Cardiac disorders) | 4 (4)
syncope (Cardiac disorders) | 1 (1)
GI bleeding (Gastrointestinal disorders) | 1 (1)
reflux esophagitis (Gastrointestinal disorders) | 1 (1)
endocarditis (Infections and infestations) | 1 (1)
systemic inflammatory response syndrome (Infections and infestations) | 1 (1)
worsening of wound healing disorder (Infections and infestations) | 1 (1)
wound infection (Infections and infestations) | 1 (1)
bleeding (Injury, poisoning and procedural complications) | 1 (1)
loosening of wire cerclages (Injury, poisoning and procedural complications) | 1 (1)
presternal abscess (Injury, poisoning and procedural complications) | 1 (1)
lumbago (Musculoskeletal and connective tissue disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1)
bronchopulmonary infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pleuropneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
pulmonary spasticity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAART 300 Annuloplasty Device (N=49)
anemia (Blood and lymphatic system disorders) | 5 (5)
aortic insufficiency (Cardiac disorders) | 7 (7)
arrhythmia (Cardiac disorders) | 20 (23)
edema (Cardiac disorders) | 5 (5)
pericardial effusion (Cardiac disorders) | 7 (7)
syncope (Cardiac disorders) | 2 (3)
abnormal LDH value (Endocrine disorders) | 2 (2)
hyperthyreosis (Endocrine disorders) | 3 (3)
increased C-reactive protein (Infections and infestations) | 6 (6)
bleeding event (Injury, poisoning and procedural complications) | 3 (3)
sternal pain (Injury, poisoning and procedural complications) | 3 (3)
thoracic pain (Musculoskeletal and connective tissue disorders) | 2 (2)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 (14)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6)
respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication by the investigator was not allowed until completion of the trial. All proposed publications must be cleared by unanimous vote of a publication committee consisting of the sponsor and representatives of the study investigators. Publication materials must be submitted for review at least 60 day in advance of publication. The Sponsor may embargo publication for 60 additional days to allow for patent filing or may prevent publication if filling of such application would be premature.